CLINICAL TRIAL: NCT06307210
Title: Clinical Effects of Inpatient Rehabilitation in Very Old Patients With Neurological, Musculoskeletal or Geriatric Disorders
Brief Title: Is Inpatient Rehabilitation Effective for Very Old Patients?
Status: Completed | Type: Observational
Sponsor: Klinik Valens (Other)
Responsible Party: Principal Investigator, Wolfgang Schallert, Principal Investigator, Klinik Valens
Other Study IDs: coreset_2020_2022
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Activity, Motor; Elderly Patients; Musculoskeletal Diseases
MeSH Terms: conditions — Motor Activity; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- age group 75-84: Inpatient rehabilitation included physiotherapy (30-60 min, 5 times/week), strength and endurance training (30-45 min, 3-5 times/week), occupational therapy (30 min, 2-3 times/week), and neuropsychological training (30 min, 2 times/week).
  Interventions: Other: inpatient rehabilitation
- age group 85-99: Inpatient rehabilitation included physiotherapy (30-60 min, 5 times/week), strength and endurance training (30-45 min, 3-5 times/week), occupational therapy (30 min, 2-3 times/week), and neuropsychological training (30 min, 2 times/week).
  Interventions: Other: inpatient rehabilitation

INTERVENTIONS:
Other: inpatient rehabilitation — physiotherapy (strength and endurance training), occupational therapy and neuropsychological training

SUMMARY:
The goal of this retrospective longitudinal observational study is to compare the effects of physical and mental performance as well as quality of life in patients with neurological and musculoskeletal disorders.

The main question it aims to answer is: Do very old patients benefit in a similar way from inpatient rehabilitation like younger patients? Data from about 2000 patients will be retrospectively analyzed. Functional Independence Measurement (FIM), Timed Up and Go Test (TUG), EuroQol 5 Dimensions (EQ-5D) and Patient Reported Outcomes Measurement Information System (PROMIS) were recorded on admission and discharge.

Researchers will compare the age group 75 to 84 and 85 to 99 to see if physical and mental performance as well as quality of life will improve.

DETAILED DESCRIPTION:
Inpatient rehabilitation has been shown to improve exercise capacity and quality of life in patients with neurological and musculoskeletal disorders.

Rehabilitation in Valens includes intensive strength and endurance training. Expectedly improvements in physical and mental performance measured by Functional Independence Measurement (FIM), Timed Up and Go Test (TUG), EuroQol 5 Dimensions (EQ-5D) and Patient Reported Outcomes Measurement Information System (PROMIS) is recognized after inpatient rehabilitation. But is this clinical effect in the same way represented in very old patients?

To the knowledge of the investigators only few studies evaluated changes after rehabilitation in patients with neurological and musculoskeletal disorders in very old patients.

Therefore, the primary goal of this study is to evaluate changes in physical and mental performance in patients with neurological and musculoskeletal disorders after inpatient rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* german speaking
* age >74
* patients with neurological and musculoskeletal disorders

Exclusion Criteria:

* age <75
* patients with pulmonological and internal disorders

Ages: 75 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Eligible subjects were German-speaking and over 74 years old referred to the Rehabilitation Centre Valens in Switzerland for inpatient rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 2270 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
FIM | 2 years
  Functional Independence Measurement; 18 categories, focusing on motor and cognitive function; each category or item is rated on a 7-point scale (1 = <25% independence; total assistance required, 7 = 100% independence); interval scale
TUG | 2 years
  Timed Up and Go Test; used to assess a person's mobility; It uses the time (in seconds) that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees; the faster the better; interval scale
EQ-5D (Quality of life) | 2 years
  EQ-5D is a standardised measure of health-related quality of life developed by the EuroQol; EQ-5D assesses health status in terms of five dimensions of health (mobility, self care, usual activities, pain and discomfort, anxiety and depression); EQ-5D is not an abbreviation and is the correct term to use when referring to the instrument; the higher the better; minimum 0, maximum 100; interval scale
PROMIS | 2 years
  Patient Reported Outcomes Measurement Information System; assessing physical, mental, and social well-being from the patient perspective; we assessed physical health (5 items, 0-10) and mental health (2 items, 0-10); interval scale

CONTACTS AND LOCATIONS:
Overall Officials: Roman Gonzenbach, Dr., Study Director — Kliniken Valens
Locations (1):
- Klinik Valens, Valens, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
not yet discussed

REFERENCES:
- [Result] Maritz R, Tennant A, Fellinghauer C, Stucki G, Prodinger B. The Functional Independence Measure 18-item version can be reported as a unidimensional interval-scaled metric: Internal construct validity revisited. J Rehabil Med. 2019 Mar 13;51(3):193-200. doi: 10.2340/16501977-2525. PMID 30843597
- [Result] Devlin NJ, Brooks R. EQ-5D and the EuroQol Group: Past, Present and Future. Appl Health Econ Health Policy. 2017 Apr;15(2):127-137. doi: 10.1007/s40258-017-0310-5. PMID 28194657
- [Result] Fries JF, Witter J, Rose M, Cella D, Khanna D, Morgan-DeWitt E. Item response theory, computerized adaptive testing, and PROMIS: assessment of physical function. J Rheumatol. 2014 Jan;41(1):153-8. doi: 10.3899/jrheum.130813. Epub 2013 Nov 15. PMID 24241485
- [Result] Valet M, Lejeune T, Devis M, van Pesch V, El Sankari S, Stoquart G. Timed Up-and-Go and 2-Minute Walk Test in patients with multiple sclerosis with mild disability: reliability, responsiveness and link with perceived fatigue. Eur J Phys Rehabil Med. 2019 Aug;55(4):450-455. doi: 10.23736/S1973-9087.18.05366-2. Epub 2018 Oct 4. PMID 30311490